CLINICAL TRIAL: NCT05919550
Title: Clozapine-associated Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Clozinfection
Record Dates: First submitted 2023-04-26; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-04

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting a possible drug-induced adverse effects
  Interventions: Drug: search for a clozapine intake

INTERVENTIONS:
Drug: search for a clozapine intake — search for a clozapine intake

SUMMARY:
perform a study in VigiBase® to assess if clozapine was associated with an over-reporting of infections and to characterize those infections. The investigators also decided to assess the dose dependency associated with those infections.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 11/04/2023
* Adverse events reported were including the MedDRA terms: infections (SOC)

Exclusion Criteria:

Chronology not compatible between the drug and the toxicity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a possible drug-induced adverse effect
Sampling Method: Probability Sample
Enrollment: 26815616 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Correlation between clozapine and hinfections using a disproportionality analysis in Individual Case Reports involving at least one liable antipsychotic drug in Vigibase® | from the 01/01/1963 to the 11/04/2023

SECONDARY OUTCOMES:
investigate a potential dose-dependent effect | from the 01/01/1963 to the 11/04/2023
  A logistical regression model will be applied to search for a dose-dependant effect of infection using clozapine quartile doses.
Description of the clinical features of clozapine-related infections | from the 01/01/1963 to the 11/04/2023
  Description of age, sex, time to onset, type of infections using MedDRA

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No